CLINICAL TRIAL: NCT00846482
Title: Exploratory Study Of The ERCC-1 Gene Expression In Colorectal Cancer Cell Lines And In Patients With Colorectal Cancer
Brief Title: Exploratory Study Of The ERCC-1 Gene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Sanjay Goel, Sanjay Goel, MD, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Purpose: Basic Science
Other Study IDs: 07-10-376
Record Dates: First submitted 2008-02-21; First posted 2009-02-18 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Colorectal cancer; Oxaliplatin; ERCC-1
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resected or metastatic CRC (Experimental): All patients with advanced or stage II or III colorectal cancer being treated with oxaliplatin
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin will be administered once every 2 or 3 weeks
  Other Names: Eloxatin

SUMMARY:
This study is for patients with advanced or stage II and III colon or rectal cancer. The primary purpose of this research study is to determine if a particular protein in the patient's blood will change when they receive treatment with a drug called oxaliplatin, which is used to treat the colon or rectal cancer. This protein is called ERCC-1. It is thought that the amount of this protein in the blood could influence the manner in which the patient responds to oxaliplatin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of colorectal cancer.
* ECOG Performance Status 0-2 (Appendix A).
* Patient is a candidate for oxaliplatin based therapy either in the adjuvant or in the metastatic setting.
* Consent to donate 4 tubes of PBMC of 7 ml of blood each.
* Willing to consider additional post therapy tumor biopsy if applicable (refusal to consent is not an exclusion criteria).
* Adequate organ function as defined as:

  * Neutrophil count > 1500/μl
  * Platelets > 75,000/ μl
  * Hemoglobin > 8 g/dl
  * Bilirubin < 2.0 X upper limit of normal
  * Creatinine < 2 mg% or calculated clearance > 40 ml/mt
* The patient must have signed a consent form approved by the Albert Einstein College of Medicine Cancer Center CCI and Montefiore Medical Center IRB

Exclusion Criteria:

* No other significant underlying medical condition that will, in the opinion of the principal investigator or designees, make administration of oxaliplatin unusually hazardous, such as significant hepatic, bone marrow and/or cardiac disease, requiring active medical treatment.
* Pregnant women or women of child bearing potential not practicing birth control or sexually active males unwilling to practice contraception during the study.
* Patients undergoing major surgical procedures (they will be delayed enrollment until complete recovery from their surgery - 4 wk for major or 2 wk from minor surgery).
* Patients with grade 2 neuropathy will not be eligible for the study.
* The patient must not have received chemotherapy within 4 weeks of beginning oxaliplatin treatment. At least 6 weeks must elapse if prior therapy included mitomycin C or nitrosoureas. At least 2 weeks must have elapsed since the end of prior palliative radiation therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-02; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SANJAY GOEL, M.D., Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Montefiore Medical Center - Weiler Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York

REFERENCES:
- [Background] Rao D, Mallick AB, Augustine T, Daroqui C, Jiffry J, Merla A, Chaudhary I, Seetharam R, Sood A, Gajavelli S, Aparo S, Rajdev L, Kaubisch A, Chuy J, Negassa A, Mariadason JM, Maitra R, Goel S. Excision repair cross-complementing group-1 (ERCC1) induction kinetics and polymorphism are markers of inferior outcome in patients with colorectal cancer treated with oxaliplatin. Oncotarget. 2019 Sep 17;10(53):5510-5522. doi: 10.18632/oncotarget.27140. eCollection 2019 Sep 17. PMID 31565185

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Resected or Metastatic CRC
Started | 64
Completed | 54
Not Completed | 10

BASELINE CHARACTERISTICS:
Population: Fifty-four patients consented to the study and underwent serial blood sampling. Blood samples were collected from every patient for at least at two of the four prespecified time points.
Arm/Group | Resected or Metastatic CRC
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 59 [45 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10
  Black | 14
  Hispanic | 26
  Asian | 2
  Unkown | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Excision Repair Cross-complementing Group-1 (ERCC1) Protein Change When Treated With Oxaliplatin
Description: ERCC was measured at the expression level, by RT-PCR and Western Blotting from peripheral blood mononuclear cells
Time Frame: Change over 1 treatment cycle, up to 4 weeks
Population: Any patient with CRC who received oxaliplatin
Measure: Count of Participants; unit: Participants
Groups:
- All Patients With CRC: All patients with advanced or stage II or III colorectal cancer being treated with oxaliplatin
  Oxaliplatin: Oxaliplatin will be administered once every 2 or 3 weeks
Arm/Group | All Patients With CRC
Number analyzed (Participants) | 50
Participants | 25

2. Secondary Outcome: Determine Extent of ERCC Polymorphism and Its Relationship to Change in Its Level
Time Frame: Change over 1 treatment cycle, up to 4 weeks
Measure: Number; unit: participants
Arm/Group | Resected or Metastatic CRC
Number analyzed (Participants) | 50
participants
  CC genotype | 22
  C/T genotype | 21
  TT genotype | 7

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | Resected or Metastatic CRC
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT00846482/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT00846482/ICF_001.pdf